CLINICAL TRIAL: NCT00720824
Title: Reduction of Immunization Discomfort in 4-6 Year Old Children: A Randomized Clinical Trial.
Brief Title: Reduction of Immunization Discomfort in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berberich, F. Ralph, M.D. (Individual)
Responsible Party: F. Ralph Berberich, MD, F. Ralph Berberich, MD
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Berberich
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2008-07-23 (Estimated); Status verified 2008-07

CONDITIONS: Pain
Keywords: Immunizations; Children; Injections; aged 4-6 Years; Hypnosis
MeSH Terms: conditions — Pain | interventions — Anesthetics, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Ethyl chloride spray, plastic arm gripper, vibrating instrument, hypnotic suggestions
  Interventions: Behavioral: Topical anesthetic and hypnotic distraction
- 2 (Placebo Comparator): Office routine
  Interventions: Behavioral: Office routine

INTERVENTIONS:
Behavioral: Topical anesthetic and hypnotic distraction — Ethyl chloride spray, plastic arm gripper, vibrating instrument, hypnotic suggestions.
  Other Names: Wahl vibrator
  Arms: 1
Behavioral: Office routine — Standard vaccine administration
  Arms: 2

SUMMARY:
A combination of topical anesthetic, plastic arm gripper, visual focusing task and hypnotic suggestions will reduce the discomfort associated with immunization of pre-kindergarten aged children.

DETAILED DESCRIPTION:
Randomization of 42 children evaluated the method described above against an office routine control group.

ELIGIBILITY:
Inclusion Criteria:

* All children ages 4-6 years scheduled to receive routine pre-kindergarten immunizations

Exclusion Criteria:

* Inability to follow verbal directions
* Significant concurrent illness
* Prior invasive procedures, excluding neonatal circumcision

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2007-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Facial Pain Scale and Faces-Legs-Activity-Cry-Consolability Scale measurements of degree of discomfort. | 10 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: f. Ralph berberich, MD, Principal Investigator — Pediatric Medial Group
Locations (1):
- Pediatric Medical Group, Berkeley, California, United States